CLINICAL TRIAL: NCT00458562
Title: HIV-Associated DNA Hypermethylation in Cervical Cancer
Brief Title: Identifying Genes That Predict Risk of Developing Cervical Intraepithelial Neoplasia or Invasive Cervical Cancer
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 6113; R01CA111187 (NIH); P30CA015704 (NIH); UWCC-6113 (Other: Fred Hutchinson/University of Washington Cancer Consortium); UWCC-04-4928-B01 (Other: Fred Hutchinson/University of Washington Cancer Consortium); FHCRC-6113 (Other: Fred Hutchinson/University of Washington Cancer Consortium); CDR0000482330 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; atypical squamous cells of undetermined significance; stage 0 cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Atypical Squamous Cells of the Cervix; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical brush in PreservCyt, cervical swab in STM, cervical swab in Roche media, whole blood, void urine, cervical tissue biopsy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV+, <CIN2: HIV positive women without CIN2-3 or worse
- HIV-, no >=CIN3 biopsy, HR HPV+: HIV negative women without biopsy-proven CIN3 or worse, and with high risk HPV infection
- HIV-, <=CIN1, HPV- at screening: HIV negative women who are <= CIN1 and HPV negative at screening

SUMMARY:
RATIONALE: Finding certain changes in genes may help doctors predict which patients are at risk of developing cervical intraepithelial neoplasia or invasive cervical cancer and may help the study of cancer in the future.

PURPOSE: This clinical trial is studying genes that may predict which patients are at risk of developing cervical intraepithelial neoplasia or invasive cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Utilize molecular assays to identify a panel of hypermethylated genes that are predictive of cervical intraepithelial neoplasia (CIN) grade 3 or invasive cervical cancer (ICC) among patients with or without HIV infection.
* Perform a nested case-control study assessing the risk of developing CIN3 in relationship to human papillomavirus (HPV) persistence, HIV, and the presence or acquisition of candidate hypermethylated genes in these patients.
* Identify HIV-related factors (e.g., CD4 counts, viral load, and highly active antiretroviral therapy [HAART]) that might be associated with the presence or acquisition of specific hypermethylated genes in these patients.

OUTLINE: This is a longitudinal, multicenter study.

Patients undergo biopsy for removal of cervical tissue. Patients also undergo blood and urine sample collection. Samples are analyzed for the presence of cancer or changes that indicate that cancer might develop. Patients also undergo colposcopy at baseline and at 3 years.

After completion of study procedures, patients are followed every 4 months for up to 3 years.

PROJECTED ACCRUAL: A total of 1,150 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Underwent Pap smear, human papillomavirus (HPV) testing, and HIV testing AND meets any of the following criteria:

  * Biopsy and colposcopy confirmed cervical intraepithelial neoplasia (CIN) or invasive cervical cancer (ICC), meeting any of the following criteria:

    * CIN grade 2-3 or higher
    * Repeated CIN1 (times 6)
    * Abnormal Pap smear (atypical squamous cells of undetermined significance [ASCUS] or worse)
  * HIV seropositive
  * Negative cytology but positive for high-risk human papillomavirus (HPV)
  * Negative cytology and negative HPV
  * HIV negative (without biopsy-proven CIN 3 or worse) and high-risk HPV infection (types 16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 55, 56, 58, 59, 68, 82, 83, 73)
* >= 18 years of age
* Intact cervix
* Not pregnant
* Able to provide informed consent

EXCLUSION CRITERIA:

* < 18 years of age
* Pregnant at screening
* Cervix not intact
* not able to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants will be African women presenting to the clinical sites in Dakar, Senegal. Subjects will be representative of ethnic and racial groups living in Senegal.
Sampling Method: Non-Probability Sample
Enrollment: 1680 (Actual)
Dates: Start 2006-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Identification of hypermethylated genes that are predictive of cervical intraepithelial neoplasia (CIN) grade 3 or invasive cervical cancer | 3 years
  Use molecular assays to identify a panel of hypermethylated genes that are predictive of CIN-3/ICC among women with and without HIV infection. We will rank genes by their ability to discriminate normal cervical tissue from CIN-3/ICC after stratifying by HIV infection.
Assessment of the risk of developing CIN3 in relationship to human papillomavirus (HPV) persistence, HIV, and the presence or acquisition of candidate hypermethylated genes | 3 years
  Perform a nested case control study assessing the risk of developing CIN-3 in relationship to HPV persistence, HIV, and the presence or acquisition of the candidate hypermethylated genes.
Identification of HIV-related factors associated with the presence or acquisition of specific hypermethylated genes | 3 years
  Identify HIV-related factors (CD4 counts, viral load, HAART) which might be associated with the presence or acquisition of specific hypermethylated genes.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy B. Kiviat, MD, Principal Investigator — Harborview Injury Prevention and Research Center
Locations (2):
- Senegal (2):
  - Centre Hospitalier Universite De Fann, Dakar
  - Hopital Aristide Le Dantec, Dakar